

# STATISTICAL ANALYSIS PLAN

### **PROTOCOL 1002-046**

A RANDOMIZED, DOUBLE-BLIND, PARALLEL GROUP, MULTICENTER STUDY
TO EVALUATE THE EFFICACY AND SAFETY OF BEMPEDOIC ACID (ETC-1002)
180 MG COMPARED TO PLACEBO ADDED TO BACKGROUND LIPIDMODIFYING THERAPY IN PATIENTS WITH ELEVATED LDL-C WHO ARE STATIN
INTOLERANT

| AUTHOR: |
|---------|

VERSION NUMBER AND DATE: V1.7, 21MAR2018

NCT number: NCT02988115
This NCT number has been applied to the document for purposes of posting on clinicaltrials.gov




### STATISTICAL ANALYSIS PLAN SIGNATURE PAGE

Statistical Analysis Plan V1.6 (Dated 14Mar2018) for Protocol 1002-046.



Upon review of this document, the undersigned approves this version of the Statistical Analysis Plan, authorizing that the content is acceptable for the reporting of this study.



Version Number: Version Date: 1.6 14Mar2018



# **MODIFICATION HISTORY**

| Unique<br>Identifier<br>for this<br>Version | Date of the<br>Document<br>Version | Author | Significant Changes from<br>Previous Authorized Version |
|---|---|---|---|
| 1.0 | 07FEB2017 | | Not Applicable – First Version |
| 1.1 | 07MAR2017 | | Changes requested from client, first review. Added appendices for multiple imputation method, AESIs and list of TLF for DMC. |
| 1.2 | 14APR2017 | | Changes requested from client, second review. |
| 1.3 | 24MAY2017 | | Changes requested from client, added new tables. |
| 1.4 | 100CT2017 | | Make relevant changes from reviews of 047 and 048 SAPs and shells. |
| 1.5 | 7JAN2018-<br>28FEB2018 | | Make Esperion's changes resulting from review of 048 dry run and 046 dry run of TLF. |
| 1.6 | 14MAR2018 | | Final changes from Esperion |
| 1.7 | 21MAR2018 | Add additional analysis for hsCRP | |

Version Number: 1.7



# **TABLE OF CONTENTS**

| | 1. | INTRODUCTION11 |
|-----|----|--------------------------------------------------------|
| | 2. | STUDY OBJECTIVES11 |
| 2.1 | | Primary Objective |
| 2.2 | | Secondary Objectives |
| 2.3 | • | Tertiary Objective |
| | 3. | STUDY DESIGN12 |
| 3.1 | | General Description |
| 3.2 | • | Schedule of Events |
| | 4. | PLANNED ANALYSES |
| 4.1 | | Data Monitoring Committee (DMC) |
| 4.2 | • | Final Analysis |
| | 5. | ANALYSIS SETS |
| 5.1 | | Safety Analysis Set [SAF] |
| 5.2 | | Full Analysis Set [FAS] |
| 5.3 | • | Completer Analysis Set [CAS] |
| 5.4 | | PK Analysis Set [PKS] |
| | 6. | GENERAL CONSIDERATIONS |
| 6.1 | | Reference Start Date and Study Day14 |
| 6.2 | • | Baseline |
| 6.3 | | Retests, Unscheduled Visits and Early Termination Data |



| 6.4. | | Visit Windowing15 |
|---|---|---|
| 6.5. | | Statistical Tests |
| 6.6. | | Common Calculations |
| <b>6.7</b> . | | Software Version |
| | <b>7</b> . | STATISTICAL CONSIDERATIONS16 |
| 7.1. | | Sample Size |
| 7.2. | | Adjustments for Covariates and Factors to be Included in Analyses |
| 7.3. | | Multicenter Studies |
| 7.4. | | Missing data |
| 7.5. | | Multiple Comparisons/ Multiplicity |
| | 8. | OUTPUT PRESENTATIONS |
| | 9. | DISPOSITION AND WITHDRAWALS |
| | <b>1</b> 1 | 1. DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS18 |
| 11.1 | | Derivations19 |
| | 12 | 2. MEDICAL AND SURGICAL HISTORY19 |
| | 13 | 3. CONCOMITANT ILLNESSES |
| | 14 | 4. CARDIOVASCULAR HISTORY/RISK FACTORS19 |
| | 15 | 5. MEDICATIONS20 |
| 15.1 | | Baseline Background Lipid Modifying Therapy20 |
| | 1 <i>6</i><br>TI | 6. ADDITIONAL POST-RANDOMIZATION ADJUNCTIVE LIPID-LOWERING HERAPY20 |

Version Number: 1.7 Version Date:

21Mar2018



| <b>17</b> . | STUDY MEDICATION COMPLIANCE AND EXPOSURE | 21 |
|---|---|---|
| 17.1. | Derivations | 21 |
| 18. | EFFICACY OUTCOMES | 22 |
| 18.1. | Primary Efficacy | 22 |
| 18.1.1 | . Primary Efficacy Variable & Derivation | 22 |
| 18.1.2 | Primary Analysis of Primary Efficacy Variable | 22 |
| 18.1.3 | Missing Data Methods for Primary Efficacy Variable | 23 |
| 18.2. | Secondary Efficacy | |
| 18.2.1 | Key secondary Efficacy Variables & Derivations | 24 |
| 18.2.2 | | |
| 18.2.3 | | |
| 18.2 | 2.3.1. Completer Analysis | |
| 18.2 | 2.3.2. Adjunctive Lipid-modifying Therapy (LMT) Analysis | |
| | 2.3.3. On-treatment Analysis | |
| | 2.3.4. Observed Data Analysis | |
| 18.2.4 | Subgroup Analysis of Efficacy Variable | 25 |
| 18.3. | Tertiary Efficacy | |
| 18.3.1 | | |
| 18.3.2 | O | |
| 18.3.3 | . 1 | |
| 18.3.4 | Additional analysis | 26 |
| 19. | SAFETY OUTCOMES | 27 |
| 19.1. | Adverse Events | 27 |
| 19.1.1 | . All TEAEs | 27 |
| 19.1 | 1.1.1. Severity | 27 |
| 19.1 | 1.1.2. Relationship to Study Medication | 27 |
| 19.1.2 | TEAEs Leading to Discontinuation of Study Medication | 28 |
| 19.1.3 | Serious Adverse Events | 28 |
| 19.1.4 | Adverse Events Of Special Interest (AESI) | 28 |
| 19.1.5 | Muscle Related Adverse Events | 28 |
| 19.2. | Deaths | 28 |
| 19.3. | Clinical Endpoints | 29 |
| 19.4. | Laboratory Evaluations | 29 |
| 19.4.1 | Laboratory Reference Ranges and Markedly Abnormal Criteria | 30 |
| 19.5. | FCG Evaluations | 31 |





| 19.6. \ | /ital Signs | 31 |
|---------|-----------------------------------------------------|----|
| 19.6.1. | Vital Signs Specific Derivations | 31 |
| 19.7. F | Physical Examination | 31 |
| 19.8. F | Pharmacokinetics | 31 |
| 20. | DATA NOT SUMMARIZED OR PRESENTED | 32 |
| 21. | REFERENCES | 32 |
| APPI | ENDIX 1.PROGRAMMING CONVENTIONS FOR OUTPUT | 33 |
| APPI | ENDIX 2.PARTIAL DATE CONVENTIONS | 40 |
| APPI | ENDIX 3.LIST OF DMC TABLES, LISTINGS AND FIGURES | 43 |
| APPI | ENDIX 4.DETAILS OF MULTIPLE IMPUTATION METHOD | 45 |
| APPI | ENDIX 5. LIST OF ADVERSE EVENTS OF SPECIAL INTEREST | 46 |

Version Number:

Version Date: 21Mar2018

1.7



### LIST OF ABBREVIATIONS

ADaM Analysis Data Model

AE Adverse Event

AESI Adverse Event of Special Interest

ANCOVA Analysis of Covariance

apoB Apolipoprotein B

ATC Anatomical Therapeutic Chemical

BLQ Below Limit of Quantification

Bpm Beats per Minute

C Celcius

CAS Completer Analysis Set

CEC Clinical Endpoints Committee

CI Confidence Interval

cm Centimeters

CV Cardiovascular; coefficient of variation

CVD Cardiovascular Disease

DBP Diastolic Blood Pressure

dL Deciliters

DMC Data Monitoring Committee

ECG Electrocardiogram

eCRF Electronic Case Report Form

eGFR Estimated Glomerular Filtration Rate

FAS Full Analysis Set

HDL-C High-density Lipoprotein – Calculated

HR Heart Rate

hsCRP High-sensitivity C-reactive Protein

IMP Investigational Medicinal Product

ITT Intention-to-treat




### LIST OF ABBREVIATIONS (cont'd)

kg kilograms

LDL-C Low-density Lipoprotein – Calculated

LDL-M Low-density Lipoprotein - Measured

LMT Lipid-modifying Therapy

LSM Least Squares Mean

LTFU Lost to Follow-up

m Meters

MACE Major Adverse Cardiac Events

MedDRA Medical Dictionary for Regulatory Activities

mg Milligrams

MI Myocardial Infarction

min Minutes

PK Pharmacokinetics

PMM Pattern Mixture Model

PT Preferred Term

SAF Safety Analysis Set

SAP Statistical Analysis Plan

SD Standard Deviation

SE Standard Error

SBP Systolic Blood Pressure

SI Systeme International

SOC System Organ Class

STDM Study Data Tabulation Model

TC Total Cholesterol

TEAE Treatment-emergent Adverse Event






### LIST OF ABBREVIATIONS (cont'd)

TG Triglycerides

ULN Upper Limit of Normal

ULQ Upper Limit of Quantification

US United States

WHO-DDE World Health Organization – Drug Dictionary Enhanced

Yrs Years




### 1. Introduction

This document describes the rules and conventions to be used in the presentation and analysis of efficacy and safety data for Protocol 1002-046. It describes the data to be summarized and analyzed, including specifics of the statistical analyses to be performed.

This statistical analysis plan (SAP) is based on the original protocol version dated August 25, 2016 and amendment 1 dated March 27, 2017.

### 2. STUDY OBJECTIVES

### 2.1. PRIMARY OBJECTIVE

The primary objective is to assess the 12-week efficacy of bempedoic acid 180 mg/day versus placebo in decreasing low-density lipoprotein cholesterol (LDL-C) in statin intolerant patients with elevated LDL-C.

### 2.2. SECONDARY OBJECTIVES

The secondary objectives are:

- To evaluate the effect of 24-week treatment with bempedoic acid 180 mg/day versus placebo on LDL-C.
- To evaluate the effect of bempedoic acid 180 mg/day versus placebo on non-high-density lipoprotein cholesterol (non-HDL-C), total cholesterol (TC), high-sensitivity C-reactive protein (hs-CRP), and apolipoprotein B (apoB) after 12 weeks of treatment.
- To evaluate the 24-week safety and tolerability of bempedoic acid 180 mg/day compared to placebo.

### 2.3. TERTIARY OBJECTIVE



### 3. STUDY DESIGN

### 3.1. GENERAL DESCRIPTION

This is a Phase 3, randomized, double-blind, placebo-controlled, parallel group multicenter study that will be conducted at approximately 71 clinical sites in North America. Screening Week -5 (Visit S1) will be approximately 5 weeks prior to randomization. Eligible patients will return to the clinical site at Week -4 (Visit S2) to initiate administration of single-blind (patient only) placebo study drug. Eligible patients will return at Week -1 (Visit S3) for lipid and safety laboratories and an assessment of tolerability and study drug adherence. Approximately 300 patients with a history of statin intolerance (SI) will be stratified based on patient type (primary prevention; secondary prevention) and randomized at Week 0 (Visit T1) in a 2:1 ratio to receive either bempedoic acid 180 mg (n = 200) or matching placebo (n = 100) once daily for 24 weeks. Randomized patients will return for clinic visits at Week 4 (Visit T2), Week 12 (Visit T4), and Week 24 (Visit T5). A phone visit will occur at Week 8 (Visit T3).

Primary and Secondary Prevention Patients with Elevated LDL-C and Statin Intolerance Bempedoic Acid 180 mg (n=200) N=300 Placebo (n=100) **Study Phase** Screen Placebo 24-Week Treatment Period Period run-in Week -5 8 12 \_1 0 4 24 Study Visit **S1** S2 T4 S3 T1 T2 T3 **T5** (phone)

Figure A 1002-046 Study Design

### 3.2. SCHEDULE OF EVENTS

The schedule of events can be found in Section 8.3 of the protocol.



### 4. PLANNED ANALYSES

The following analyses will be performed for this study:

- Safety analyses for Data Monitoring Committee (DMC) meetings
- Final Analysis

## 4.1. DATA MONITORING COMMITTEE (DMC)

The subset of outputs for the DMC is listed in Appendix 3. Access to results will be provided by Quintiles in a separate unblinding plan.

### 4.2. FINAL ANALYSIS

All final, planned analyses identified in this SAP will be performed by Quintiles Biostatistics following Sponsor Authorization of this Statistical Analysis Plan, Database Lock, Sponsor Authorization of Analysis Sets and Unblinding of Treatment.

### 5. ANALYSIS SETS

Agreement and authorization of subjects included/ excluded from each analysis set will be conducted prior to the unblinding of the study.

# 5.1. SAFETY ANALYSIS SET [SAF]

The Safety Analysis Set (SAF), used for all of the safety summaries, is defined as all randomized patients who received at least 1 dose of double-blind study medication. Patients in the SAF will be included in the treatment group that they actually received, regardless of their randomized treatment.

# 5.2. FULL ANALYSIS SET [FAS]

The Full Analysis Set (FAS), used for all of the efficacy analyses, is defined as all randomized patients. The FAS is also known as the intention-to-treat (ITT) set of patients. Patients in the FAS will be included in their randomized treatment group, regardless of the treatment they actually received.



## 5.3. COMPLETER ANALYSIS SET [CAS]

The Completer Analysis Set (CAS), used for all the primary, and secondary efficacy analysis, is defined as patients who completed IMP treatment per the end of treatment CRF page and have non-missing week 12 LDL-C value.

## 5.4. PK ANALYSIS SET [PKS]

The PK Analysis Set will include all subjects in the safety analysis set who have at least one non-missing PK assessment. These subjects will be evaluated for PK concentration summaries unless major protocol deviations are identified during the protocol deviation review or if key dosing or sampling information is missing.

### 6. GENERAL CONSIDERATIONS

### 6.1. REFERENCE START DATE AND STUDY DAY

Study Day will be calculated from the reference start date, and will be used to show start/ stop day of assessments and events.

Reference start date is defined as the day of the first dose of study medication (Day 1 is the day of the first dose of study medication). In case the first dose date is missing, randomization date will be used instead.

If the date of the event is on or after the reference date then:

Study Day = (date of event - reference date) + 1.

If the date of the event is prior to the reference date then:

Study Day = (date of event – reference date).

In the situation where the event date is partial or missing, the date will appear partial or missing in the listings, and Study Day, and any corresponding durations will be presented based on the imputations specified in Appendix 2: Partial Date Conventions.

### 6.2. BASELINE

Unless otherwise specified, baseline is defined as the last non-missing measurement taken prior to



reference start date (including unscheduled assessments). In the case where the last non-missing measurement and the reference start date coincide, that measurement will be considered as baseline, but Adverse Events (AEs) and medications commencing on the reference start date will be considered post-baseline.

Baseline for calculated LDL-C, non-HDL-C, and TC is defined as the mean of the values from Week -1 (Visit S3) and predose Day 1/Week 0 (Visit T1) (i.e., the last two non-missing values on or prior to Day 1). If only one value is available then that single value will be used as baseline.

Baseline for apoB and hs-CRP is defined as the predose Day 1/Week 0 (Visit T1) value (i.e. the last non-missing value on or prior to Day 1). If this is not available, then the last non-missing value prior to the first dose of double-blind study medication (including unscheduled assessments) will be used as baseline.

### 6.3. RETESTS, UNSCHEDULED VISITS AND EARLY TERMINATION DATA

In the event of a missing value at a scheduled visit, and if an unscheduled visit falls within the protocoldefined window of that visit (see table below), the value from the unscheduled visit will be used for that visit.

In the case of a retest (same visit number assigned), the later available measurement for that visit will be used for by-visit summaries.

Listings will include scheduled, unscheduled, retest and early discontinuation data.

### 6.4. VISIT WINDOWING

Protocol-defined assessments will be "slotted" to study weeks based on collection date and applying the rules summarized in the following table. If there is more than one scheduled visit in a visit window, the visit closest to the target date will be used. If there is a tie between the numbers of days from the target date, the visit after the target date will be used. Unscheduled visits that fall within the protocol-defined visit windows will be summarized in the by-visit analyses if there is no scheduled visit available. If there is more than one unscheduled visit within the protocol-defined visit window and no scheduled visit available, the unscheduled visit closest to the scheduled visit date will be used. If there is a tie between the numbers of days from the target date, the visit after the target date will be used.

However, exposure data obtained from the drug accountability and administration CRF will be summarized and listed according to nominal visit information

| Visit | S1 | S2 | S3 | T1 | T2 | T3 | T4 | T5, EOS |
|---------------------------|-----|-----|----|----|----|----|----|---------|
| <b>Slotted Study Week</b> | -5 | -4 | -1 | 0 | 4 | 8 | 12 | 24 |
| Target Study Day | -35 | -28 | -7 | 1 | 29 | 57 | 85 | 168 |



### 6.5. STATISTICAL TESTS

The default significance level will be (5%); confidence intervals will be 95% and all tests will be two-sided, unless otherwise specified in the description of the analyses.

### 6.6. COMMON CALCULATIONS

For quantitative measurements, change from baseline will be calculated as:

Test Value at Visit X – Baseline Value

Percent change from baseline will be calculated as:

• [(Test Value at Visit X – Baseline Value)/Baseline Value] x 100

### **6.7. SOFTWARE VERSION**

All analyses will be conducted using SAS version 9.4 or higher.

### 7. STATISTICAL CONSIDERATIONS

### 7.1. SAMPLE SIZE

The primary efficacy endpoint for this study is the percent change from baseline to Week 12 in LDL-C.






# 7.2. ADJUSTMENTS FOR COVARIATES AND FACTORS TO BE INCLUDED IN ANALYSES

The following covariates and factors are used in the analyses. For details of their inclusion in the models, see the specific analysis section.

- treatment group (bempedoic acid 180 mg/day; placebo)
- baseline laboratory value of interest
- CVD risk category (primary prevention; secondary prevention)
- treatment by subgroup interaction term for subgroup analyses of efficacy variables

### 7.3. MULTICENTER STUDIES

This study will be conducted by multiple investigators at multiple centers in North America.

### 7.4. Missing data

Missing efficacy data will be handled as described in section 18.1.2 of this analysis plan.

## 7.5. MULTIPLE COMPARISONS/ MULTIPLICITY

In terms of controlling the overall Type I error rate, a gatekeeping or stepdown approach will be used to test the primary efficacy endpoint and then specific secondary efficacy endpoints sequentially in order to preserve the study-wise Type I error rate. The sequence for the stepdown procedure in this study is as follows:

- 1. Test the primary efficacy endpoint: percent change from baseline to Week 12 in LDL-C
- 2. Test the percent change from baseline to Week 24 in LDL-C
- 3. Test the percent change from baseline to Week 12 in non-HDL-C
- 4. Test the percent change from baseline to Week 12 in TC
- 5. Test the percent change from baseline to Week 12 in apoB
- 6. Test the percent change from baseline to Week 12 in hsCRP

In this hierarchical testing structure, each hypothesis is tested at a significance level of 0.05, twosided. Statistical significance at each step is required in order to test the next hypothesis. If the primary endpoint meets the criteria for statistical significance, then the percent change from



baseline to Week 24 in LDL-C will be tested; and so forth.

### 8. OUTPUT PRESENTATIONS

Appendix 1 shows conventions for presentation of data in outputs.

The templates provided with this SAP describe the presentations for this study and therefore the format and content of the summary tables, figures and listings to be provided by Biostatistics.

### 9. DISPOSITION AND WITHDRAWALS

All patients who were screened will be accounted for in this study. Reasons for screen failure will be summarized by pre-defined categories per CRF. For screen failure due to inclusion and exclusion criteria, the criteria category will be presented. Patient disposition and withdrawals (both from study treatment and the study), will be presented for the FAS. The number of patients in each analysis set will be presented for all randomized patients.

### 10. PROTOCOL DEVIATIONS

All protocol deviations will be provided in a listing with type and description. Major protocol deviations will be summarized by treatment group. The protocol deviations are recorded and tracked in the trial monitoring platform CTMS.

### 11. Demographic and other Baseline Characteristics

Demographic data and other baseline characteristics will be presented for the FAS and CAS. No statistical testing will be carried out for demographic or other baseline characteristics. The following demographic and other baseline characteristics will be reported for this study:

- Age (years) calculated relative to date of randomization
- Age category (<65 years vs. ≥65 years and < 75 years vs. ≥75 years)</li>
- Gender
- Race
- Ethnicity
- CVD risk category (primary prevention; secondary prevention)
- Region (US vs. Canada)
- Weight (kg)
- Height (cm)

Version Date: 21Mar2018




- BMI (kg/m2)
- BMI category (< 25 vs. 25 < 30 vs. ≥ 30 kg/ m2)
- Baseline Laboratory Results (Total Cholesterol, LDL-C, HDL-C, Triglycerides, Non-HDL-C, ApoB, and hsCRP)
- Baseline LDL-C category (<130 mg/dL, ≥130 and < 160 mg/dL, or ≥160 mg/dL)</li>
- Background lipid modifying therapy use (Statin vs. Non-statin vs. None)
- History of diabetes (Yes vs. No)
- History of hypertension (Yes vs. No)
- Baseline Vital Signs (systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR)
- Alcohol consumption
- Tobacco use

### 11.1. DERIVATIONS

- Age (years) = (date of randomization date of birth)/365.25
- BMI (kg/m2) = weight (kg)/ height (m)2

### 12. MEDICAL AND SURGICAL HISTORY

Medical and Surgical History information will be presented by MedDRA SOC (System Organ Class) and PT (Preferred Term) for the FAS. Medical History conditions are defined as those conditions which stopped prior to or at Screening. Medical and Surgical History will be coded using MedDRA Version 20.1.

### 13. CONCOMITANT ILLNESSES

Concomitant Illnesses will be presented by SOC (System Organ Class) and PT (Preferred Term) for the FAS. Concomitant Illnesses are conditions (other than the indication being studied) which started prior to the date of randomization and are ongoing at the date of randomization. Concomitant Illnesses will be coded using MedDRA Version 20.1.

## 14. CARDIOVASCULAR HISTORY/RISK FACTORS

Cardiovascular history/risk factors collected at screening will be presented in a table by treatment group and in a data listing.




### 15. MEDICATIONS

Prior and concomitant medications will be presented for the SAF and coded using the September 2017 version of the World Health Organization Drug Dictionary Enhanced (WHO-DDE). Tables excluding lipid-modifying therapies will be presented.

Prior and concomitant lipid modifying therapy including statin (less than low dose) and others will be tabulated and listed separately. See protocol section 7.3.1 for the list of LMT allowed in the study.

Medications will be summarized by ATC classification and preferred term by treatment group.

See Appendix 2 for handling of partial dates for medications, in the case where it is not possible to define a medication as prior or concomitant to treatment, the medication will be classified by the worst case, i.e. concomitant.

Prior medications are medications which started and stopped prior to the first dose of double-blind study medication.

Concomitant medications are medications that patients are taking at the time of first dose of double-blind medication or started during the study, which means: started prior to, on or after the first dose of double-blind study medication and no later than 30 days following the end of study medication, and ended on or after the date of first dose of study medication or were ongoing at the end of the study.

### 15.1. BASELINE BACKGROUND LIPID MODIFYING THERAPY

Baseline background Lipid modifying therapy is defined as any lipid modifying agents that are ongoing at the time of randomization. It will be presented in separate tables and listings by category (as defined in protocol section 7.3.1) and coded medication name and by treatment group.

### 16. Additional Post-randomization Adjunctive Lipid-Lowering Therapy

The number and percent of patients in each treatment group requiring additional (post-randomization) lipid-lowering therapy will be summarized by treatment group as well as provided in a listing. The lipid-lowering therapy includes all post-randomization concomitant medications based on ATC class 2 = lipid-modifying agent.



### 17. STUDY MEDICATION COMPLIANCE AND EXPOSURE

Compliance to study medication will be presented for the SAF. At visits Week -1 (S1), Week 0 (T1), and each patient visit during the study, clinical site staff will count the number of tablets that are returned as unused and query the patient with regards to daily intake.

### 17.1. DERIVATIONS

Compliance with placebo-run in (as an overall group) and double-blind study medication by treatment group—based on the drug accountability data—will be calculated as the number of tablets taken (total dispensed – total returned) divided by the number of days on treatment within each of the 2 periods.

During the run-in period, the compliance will be summarized as a single overall group and during the double-blind period, compliance will be summarized by treatment group (bempedoic acid and placebo).

Compliance will not be computed by visit.

A 35-day supply of single-blind placebo drug will be dispensed one time at Week -4 (Visit S2) for the 4-week placebo run-in period of the study. Double-blind IMP will be dispensed in 100 day supply increments to patients by appropriate clinical site personnel. Patients will receive one 100-day supply bottle at Week 0 (Visit T1)).

The treatment is taken once daily and it is assumed that the patient takes medication on the visit day at which their medication is initially dispensed to the date of last dose as captured on the End of Treatment eCRF page. For example, if the initial dispense date is Day 1 and the last dose is Day 84, then the patient should have taken the first tablet at Day 1, once a day on Days 2 to 83 and 1 tablet on Day 84; hence, the total number of prescribed tablets would be 84.

For subjects who did not return any bottle during the double-blind period, their compliance will be set to missing.

Treatment exposure will be calculated in weeks as (date of last dose of study medication – first date of first dose of study medication +1)/7. Descriptive statistics will be presented for exposure as well as categorization into time periods (e.g., <12weeks, >=12 weeks to <24 weeks, >=24 weeks, etc.).



### 18. EFFICACY OUTCOMES

### 18.1. PRIMARY EFFICACY

### 18.1.1. PRIMARY EFFICACY VARIABLE & DERIVATION

The primary efficacy endpoint is the percent change from baseline to Week 12 in LDL-C. Baseline LDL-C is defined as the mean of the LDL-C values from Week -1 (Visit S3) and predose Day 1/Week 0 (Visit T1).

In cases where triglycerides (TG) is >400 mg/dL or LDL-C is <=50 mg/dL, a measured LDL (LDL-M) will be used instead of LDL-C for the analysis of that time point. If both values are available, the LDL-M will be used.

### 18.1.2. PRIMARY ANALYSIS OF PRIMARY EFFICACY VARIABLE

The null hypothesis, H<sub>0</sub>, will be that there is no difference between bempedoic acid 180 mg/day and placebo in mean percent change from baseline to Week 12 in LDL-C. The alternative hypothesis, H<sub>1</sub>, will be that bempedoic acid 180 mg/day is different from placebo:

 $H_0: \mu_p = \mu_b$ 

 $H_1$ :  $\mu_p \neq \mu_b$ 

where  $\mu_p$  and  $\mu_b$  denote the mean percent change from baseline to Week 12 in LDL-C on placebo and bempedoic acid 180 mg/day respectively.

The primary efficacy endpoint will be analyzed using analysis of covariance (ANCOVA), with treatment group and stratification factor patient type as factors and baseline LDL-C as a covariate. To account for the likelihood of unequal variances between the treatment groups, the ANCOVA model will be implemented within mixed model framework and the repeated/group=> option will be used to allow estimating the residual variances separately between the groups. Model assumptions for performing ANCOVA will be assessed and if the assumptions are severely violated, non-parametric methods will be performed.

In addition, descriptive statistics will be presented for LDL-C at each visit and for change from baseline and % change from baseline.





# 18.1.3. MISSING DATA METHODS FOR PRIMARY EFFICACY VARIABLE

For the primary endpoint of percent change from baseline to Week 12 in LDL-C values, a pattern mixture model (PMM) will be used to specify different imputation strategies depending on whether the patient is still on study treatment. Patients with missing lipid data at Week 12 who are no longer taking study treatment (defined by date of last dose of study medication is < Week 12 lab assessment date -7) can be assumed to no longer be benefitting from study medication, and their missing value(s) can be assumed to be similar to those in placebo group who remained on study and have data. To account for uncertainty, missing values will be imputed using multiple imputation via a regression based model including stratification and baseline data from placebo subjects only. In this imputation model, treatment group will not be included as a factor.

Patients with missing lipid data at Week 12 who are still taking study treatment (date of last dose of study medication is ≥ Week 12 lab assessment date -7) can be assumed to continue to benefit from study medication, and their missing value(s) can be assumed to be similar to those who remain on study treatment and have data and as a result, lipid values will be imputed based on the observed values in their randomized treatment group at Week 12. To account for uncertainty, missing values will be imputed using multiple imputation via a regression based model including treatment, stratification and baseline value.

Imputed datasets will be analyzed using the same ANCOVA model with treatment and stratification as factors and baseline LDL-C as a covariate descried in section 18.1.2. Approximately 200 imputed datasets will be created, with results from the analysis of each imputed dataset combined using Rubin's method. The least squares mean (LSM) and standard error (SE) will be provided for both treatment groups, along with the placebo-corrected LSM, its 95% confidence interval (CI) and associated p-value. To account for possibility of unequal variances between the groups, the ANCOVA model will be implemented within mixed model framework where <repeated/group=> option will be used to allow separate estimation of residual variance between the groups.

Further information on the multiple imputation method is presented in Appendix 4.

### 18.2. SECONDARY EFFICACY

The secondary efficacy analyses will be performed for the full analysis set (FAS).



# 18.2.1. Key secondary Efficacy Variables & Derivations

The key secondary endpoints, which are included in the hierarchical analysis described in Section 7.5, are:

- percent change from baseline to Week 24 in LDL-C
- percent change from baseline to Week 12 in non-HDL-C
- percent change from baseline to Week 12 in TC
- percent change from baseline to Week 12 in apoB
- percent change from baseline to Week 12 in hsCRP.

Key secondary endpoints of LDL-C, non-HDL-C, TC, and apoB will be analyzed using the same ANCOVA model described in 18.1.2.

Similar to the primary endpoint, missing data will be imputed using multiple imputation method as described in 18.1.3.

For hsCRP, a non-parametric (Wilcoxon rank-sum test) analysis with Hodges-Lehmann estimates and confidence interval will be performed because based on historical knowledge, publication precedence (Brendan etc., 2006) and recent data available, hsCRP is known to be skewed by extreme values and have non-normal distribution.

Graphic presentations (mean+/-SE) or median (IQR) for efficacy parameters will be provided.

# **18.2.2.** OTHER SECONDARY EFFICACY VARIABLES & DERIVATIONS

Other secondary efficacy endpoints are:

- Change from baseline to Week 12 in LDL-C
- Change from baseline to Week 24 in LDL-C.

The absolute change in LDL-C at week 12, 24 will be summarized using descriptive statistics.

# 18.2.3. SENSITIVITY ANALYSIS OF PRIMARY AND KEY SECONDARY EFFICACY VARIABLES

### 18.2.3.1. Completer Analysis

The completer analysis set (CAS) will be used as a sensitivity analysis for all primary and key secondary efficacy endpoints. There will be no imputation for missing data.




#### 18.2.3.2. Adjunctive Lipid-modifying Therapy (LMT) Analysis

To explore the potential impact from adjunctive lipid-modifying therapy use during the study, a sensitivity analysis will be performed for primary and key secondary endpoints using data prior to the change of the post-baseline LMT only, i.e., lab test date <=change date of LMT. There will be no imputation for missing data.

#### 18.2.3.3. **On-treatment Analysis**

An on-treatment analysis will also be conducted for primary and key secondary endpoints using data collected from the on-treatment period, i.e. lab test date <= of last dose of double-blind IMP+7 days. On-treatment analysis will be based on FAS. There will be no imputation for missing data.

#### 18.2.3.4. **Observed Data Analysis**

The observed case data with no imputation for missing data will be used in sensitivity analyses for primary and key secondary endpoints.

### 18.2.4. SUBGROUP ANALYSIS OF EFFICACY VARIABLE

The primary endpoint for LDL-C will be analysed within subgroups below using the same analysis method previously described. The treatment and subgroup interaction will be examined by including the interaction term in the ANCOVA model for the overall population first. No imputation will be performed on missing data for subgroup analyses. In case the number of subjects within a subgroup is too small, e.g. less than 5% of the overall population, the analyses may not be performed or the subgroup levels may be combined. Forest plots for the primary efficacy variable will also be presented.

- CVD risk category (primary prevention; secondary prevention)
- Baseline LDL category (<130mg/dL, ≥130 mg/dL and < 160 mg/dL, ≥160mg/dL)</li>
- History of diabetes (yes vs.no)
- Age (< 65 yrs. vs. ≥65 yrs. and <75 yrs vs. ≥75 yrs)</li>
- Race (White vs. Non-White))
- Gender (male vs. female)
- BMI category (< 25 vs. 25 < 30 vs.  $\geq$  30 kg/ m2)
- Background lipid modifying therapy (statin vs. non-statin vs. none)


21Mar2018 Version Date:



# 18.3. TERTIARY EFFICACY

### 18.3.1. TERTIARY EFFICACY VARIABLES & DERIVATIONS

The tertiary efficacy endpoints are:



# **18.3.2.** Missing Data Methods for Tertiary Efficacy Variables

No missing data imputation will be performed for the tertiary endpoint analyses, only observed data will be used.

### 18.3.3. ANALYSIS OF TERTIARY EFFICACY VARIABLES



18.3.4. ADDITIONAL ANALYSIS



### 19. SAFETY OUTCOMES

All outputs for safety outcomes will be based on the Safety Analysis Set.

There will be no statistical comparisons between the treatment groups for safety data, unless otherwise specified with the relevant section.

### 19.1. ADVERSE EVENTS

Adverse Events (AEs) will be coded using MedDRA, Version 20.1.

Treatment emergent adverse events (TEAEs) are defined as AEs that started or worsened in severity after the first dose of IMP (double-blind study medication) and prior to the last dose date of double-blind study medication + 30 days. AEs that occurred on day 1 will be only be determined as TEAE if the site indicated it occurred after first dose on the AE CRF.

See Appendix 2 for handling of partial dates for AEs. In the case where it is not possible to define an AE as treatment emergent or not, the AE will be classified by the worst case, i.e. treatment emergent.

An overall summary of number of subjects within each of the categories described in the subsection below, will be provided as specified in the templates. Listings will include TEAEs and Non-TEAEs.

#### 19.1.1. ALL TEAES

Incidence of TEAEs will be presented by System Organ Class (SOC) and Preferred Term (PT) and also broken down further by maximum severity and relationship to study medication. Adverse events by the subgroups in Section 18.2.4 with the exception of baseline LDL subgroup will also be presented.

### 19.1.1.1. Severity

Severity is classed as mild/ moderate/ severe (increasing severity). TEAEs starting after the first dose of IMP with a missing severity will be classified as severe. If a patient reports a TEAE more than once within that SOC/ PT, the AE with the worst case severity will be used in the corresponding severity summaries.

### 19.1.1.2. Relationship to Study Medication

Relationship to IMP, as indicated by the Investigator, is "not related" if the TEAE is "not related" or "unlikely". A "related" TEAE is defined as a TEAE with a relationship of "possibly related", "probably related", or "definitely related" to study medication. TEAEs with a missing relationship



to study medication will be regarded as "probably related" to study medication. If a patient reports the same AE more than once within that SOC/ PT, the AE with the worst case relationship to study medication will be used in the corresponding relationship summaries.

# 19.1.2. TEAES LEADING TO DISCONTINUATION OF STUDY MEDICATION

TEAEs leading to permanent discontinuation of study medication will be identified by using the response of 'Drug Withdrawn/Permanently discontinued' on the Action Taken with Study Drug Field on the AE eCRF page. For TEAEs leading to discontinuation of study medication, summaries of incidence rates (frequencies and percentages) by SOC and PT will be summarized.

### 19.1.3. SERIOUS ADVERSE EVENTS

Serious adverse events (SAEs) are those events recorded as 'serious' on the adverse events page of the eCRF. Summaries of serious TEAEs and serious related TEAEs by SOC and PT will be prepared.

### 19.1.4. ADVERSE EVENTS OF SPECIAL INTEREST (AESI)

Adverse events of special interest will be identified by pre-specified MedDRA preferred terms provided by Esperion Therapeutics Inc. (see Appendix 5). These events will be summarized by AESI category, SOC and PT. All AESI will be summarized by severity and relationship to study medication. In addition, AESI will be evaluated by monitoring safety labs as detailed in section 19.4.

### 19.1.5. Muscle Related Adverse Events

Muscle related events as reported on the general AE CRF will be summarized by maximum severity and SOC and PT. All muscle related events and details associated with it including cause and location will be provided in a listing.

### **19.2. DEATHS**

If any patient dies during the study, as recorded on the Death Event page of the eCRF, the information will be presented in a data listing. Deaths will be categorized as cardiovascular (CV) death (MACE) or non-CV death (non-MACE).



### 19.3. CLINICAL ENDPOINTS

Clinical endpoints will be monitored and adjudicated by an independent blinded expert CEC for this study. The following clinical endpoints will be tabulated:

- CV death (MACE)
- Nonfatal myocardial infarction [MI] (MACE)
- Nonfatal stroke (MACE)
- Hospitalization for unstable angina (MACE)
- Coronary revascularization (MACE)
- Non-coronary arterial revascularization (non-MACE)
- Hospitalization for heart failure (non-MACE)
- Non-CV death (non-MACE)

Additional details regarding clinical endpoints and clinical endpoint definitions will be included in CEC charter. The number of incidences and percentage of patients with each positively adjudicated outcome will be presented in a table. Only treatment emergent positively adjudicated events will be presented in the summary table. All adjudicated events will be included in a listing.

### 19.4. LABORATORY EVALUATIONS

Results from the central laboratory will be included in the reporting of this study for Hematology, Blood Chemistry, Lipids, Coagulation, HbA1c, hsCRP and Urinalysis. A list of laboratory assessments to be included in the outputs is included in Protocol, Section 10.1.6.1.

Presentations will use SI Units and conventional units.

Quantitative laboratory measurements reported as "< X", i.e. below the lower limit of quantification (BLQ), or "> X", i.e. above the upper limit of quantification (ULQ), will be converted to X for the purpose of quantitative summaries, but will be presented as recorded, i.e. as "< X" or "> X" in the listings.

The formula to calculate eGFR is: eGFR =  $186 \times (Creatinine / 88.4)-1.154 \times (Age)-0.203 \times (0.742 if female) \times (1.210 if black), where creatinine is in mmol/L.$ 

Summaries for all lab results, including unscheduled visit values, will be included for below analyses:

Observed and change/percent change from baseline by visit (for quantitative measurements).



- Observed and change/percent change from baseline for HbA1c and glucose by history of diabetes and visit.
- Shift from baseline by visit according to normal ranges.
- Shift from baseline according to normal ranges for HbA1c and glucose by history of diabetes and visit.
- eGFR and values of CK will be summarized by treatment group and by baseline eGFR categories (low, normal, high).
- Potential Hy's law cases (>3 × ULN for ALT and/or AST with concurrent Total Bilirubin >2 × ULN) will be tabulated listed.
- Laboratory abnormalities in parameters of interest

ALT or AST (> 3x ULN , >5xULN)
TB (>2x ULN)

CK (> 5x ULN) and (>10x ULN)

Fasting Blood Glucose (≤50 mg/dL, ≥126 mg/dL) by history of diabetes

HbA1c (≥6.5%) by history of diabetes

Creatinine (change from baseline for >1 mg/dL)

eGFR (< 15 mL/min/1.73m<sup>2</sup>, 15 -< 30 mL/min/1.73m<sup>2</sup>)

Hgb (decrease from baseline for ≥2 g/dL)

Hgb (<8 g/dL)

# 19.4.1. LABORATORY REFERENCE RANGES AND MARKEDLY ABNORMAL CRITERIA

Quantitative laboratory measurements will be compared with the relevant laboratory reference ranges in SI units and categorized as:

- Low: Below the lower limit of the laboratory reference range.
- Normal: Within the laboratory reference range (upper and lower limit included).
- High: Above the upper limit of the laboratory reference range.

In addition to the high and low quantitative laboratory assignments, Hy's law criteria (≥3 × ULN for either ALT or AST, with accompanying total bilirubin >2 × ULN in the absence of other known causes) will be used to identify potential Hy's law cases.




### 19.5. ECG EVALUATIONS

The Investigator's judgment of overall assessment of ECG (Normal, Abnormal, Not Clinically Significant [ANCS], and Abnormal, Clinically Significant [ACS]) will be recorded at baseline and end of study. A summary of shift from baseline to end of study in overall assessment will be provided.

### 19.6. VITAL SIGNS

The following Vital Signs measurements will be reported for this study:

- Sitting Systolic Blood Pressure (mmHg)
- Sitting Diastolic Blood Pressure (mmHg)
- Sitting Heart Rate (bpm)
- Weight (kg)
- Height (cm) (at Screening only)
- BMI (kg/m²) (calculated automatically by the EDC system)

The following summaries will be provided for vital signs data: Observed and change from baseline by visit.

### 19.6.1. VITAL SIGNS SPECIFIC DERIVATIONS

Blood pressure is taken twice five minutes apart at each vital sign collection. Blood pressure will be analyzed as the average of these two measurements. If there is only 1 measurement, that measurement will be used.

### 19.7. Physical Examination

Abnormalities in physical examinations will be presented in a listing.

### 19.8. PHARMACOKINETICS

Descriptive statistics for concentrations of bempedoic acid and its metabolite ESP15228 will be presented for each visit weeks 4, 8, and 12 if the PK sample time is within 18-30 hours of the last dose of IMP. All concentration data will also be presented in a listing. All concentrations below the limit of quantification or missing data will be labelled as such in the concentration data listings. Concentrations below the lower limit of quantification will be treated as zero in summary statistics.



### 20. DATA NOT SUMMARIZED OR PRESENTED

The other variables and/or domains not summarized or presented are:

- Comments
- Variables used by the data entry system to direct user to proper page (e.g., patient visit status, patient health status)
- Inclusion/Exclusion Criteria that are not violated
- Normal Physical Examination Results
- Diet and Exercise Counselling
- Normal PE findings

These domains and/or variables will not be summarized or presented, but will be available in the clinical study database, SDTM and/or ADaM datasets.

### 21. REFERENCES

ICH E9. E9 Statistical Principles for Clinical Trials. Federal Register. 1998; 63(179):49583-49598.

Little, R. & Rubin, D.(1987) Statistical Analysis with Missing Data, Wiley, New York.

Ratitch, B. and O'Kelley, M., "Implementation of Pattern-Mixture Models Using Standard SAS/STAT Procedures," in Proceedings of PharmaSUG 2011 (Pharmaceutical Industry SAS Users Group), SP04,

Nashville.

O'Brien, Peter C., and Thomas R. Fleming. "A multiple testing procedure for clinical trials." Biometrics (1979): 549-556.

Demets, David L., and K. K. Lan. "Interim analysis: the alpha spending function approach." Statistics in medicine 13.13-14 (1994): 1341-1352.

Brendan M.Everett, TobiasKurth, Julie E.Buring, Paul M.Ridker. "The Relative Strength of C-Reactive Protein and Lipid Levels as Determinants of Ischemic Stroke Compared With Coronary Heart Disease in Women." Journal of the American College of Cardiology (2006), Volume 48, Issue 11, Pages 2235-2242.




### **APPENDIX 1. Programming Conventions for Output**

**Quintiles Output Conventions** 

File names should only consist of uppercase letters, lowercase letters, digits (0 to 9) and underscores. A period should only be used to indicate a separator between the file name and the extension. No spaces, other special characters or punctuation marks are permitted.

As far as possible, output files should be in RTF format, although .DOC files are also permitted.

The program, program log and output file name should reflect the type and number of the statistical output. If this is not possible, then the output name should be at least as descriptive as possible. A prefix can be used to distinguish between a Table, Listing and Figure document ('T' for table, 'L' for listing and 'F' for figure). If there is only 1 digit in the number of the table, listing or figure in the place where 2 digits are possible, a leading zero should be added in the file name to make sorting consistent with the sequence (eg T14\_3\_01\_1.RTF).

### PAPER SIZE, ORIENTATION AND MARGINS

The size of paper will be Letter for the United States, otherwise A4.

The page orientation should preferably be landscape, but portrait is also permitted.

Margins should provide at least 1 inch (2.54 centimeters) of white space all around the page, regardless of the paper size.

The number of columns per page (linesize) should be 145 for A4 and 134 for Letter.

The number of rows per page (pagesize) should be 49 for A4 and 51 for Letter.



#### **FONTS**

The font type 'Courier New' should be used as a default for tables and listings, with a font size of 8. The font color should be black. No **bolding**, underlining *italics* or subscripting should be permitted. Try to avoid using super-scripts, unless absolutely necessary. Single spacing should be used for all text. Figures should have a default font of "Times Roman", "Helvetica", or "Courier New".

This can be achieved by using the following options in SAS:

```
goptions
gunit = pct
cback = white
colors = (black)
hby = 2.4
ftext = "TimesRoman"
htext = 2.5
device = cgmof97l
gaccess = gsasfile;
filename gsasfile "....cgm";
```

### **HEADER INFORMATION**

Headers should be defined as follows:

- The header should be placed at the top of the page (same place on each page) regardless of the size or orientation of the table or listing
- The customer name and protocol number should appear in row 1, left-aligned
- The output identification number should appear in row 2, centered
- The output title should start in row 3, centered
- The output population should appear in row 4, centered. The population should be spelled out in full, e.g. Intention-to-Treat in preference to ITT.
- Row 5 should be a continuous row of underscores ('\_') (the number of underscores should equal the linesize)
- Row 6 should be a blank line
- Mixed case should be used for titles
- The output titles should be designed so that they are arranged consistently through all outputs. For example, content (eg Vital Signs) followed by metric (eg Change from Baseline) e.g. Vital Signs Change from Baseline.
- Titles should not contain quotation marks or footnote references
- The column headings should be underlined with a row of underscores ('\_')
- Column headings spanning more than one column should be underlined and have underscores on either side of the title and should be centered
- Column headings containing numbers should be centered
- Column headings should be in sentence case
- In general, the population count should appear in the column header in the form "(N=XXX)"



- "Statistic" should be the column header over n, Mean, SE, n (%) etc.
- As a rule, all columns should have column headings.

#### TABLE AND LISTING OUTPUT CONVENTIONS

### General:

- The first row in the body of the table or listing should be blank
- The left hand column should start in column 1. No indenting or centering of the output should occur.
- Rounding should be done with the SAS function ROUND.
- Numbers in tables should be rounded, not truncated.
- Alphanumeric output should be left aligned.
- Numbers should be decimal point aligned.
- Whole numbers should be right aligned.
- Text values should be left aligned.
- The first letter of a text entry should be capitalized
- Listings of adverse events, concomitant medications, medical histories etc. should be sorted in chronological order, with earliest adverse event, medication or history coming first.
- The study drug should appear first in tables with treatments as columns
- In general, only present totals (across treatment groups) at baseline/randomization, and do not present them post randomization, unless the customer specifically requests it.
- If possible, include 100% frequencies in the table shell, so that it is clear what the denominator is for percentage calculations.
- All listing outputs should be sorted (preferably by Treatment, Site Number and Subject Number).
- Do not use superscripts and subscripts
- Exponentiation will be expressed using a double asterisk, i.e., mm3 will be written as mm\*\*3.
- All variables that are output in the CRF (which have data present) should appear in the listings, along with all derived data appearing in the corresponding tables
- The width of the entire output should match the linesize

### **Univariate Statistics:**

- Statistics should be presented in the same order across tables (i.e., n, Mean, SD, Q1, Median, Q3, Minimum, Maximum)
- Table statistics should line up under the N part of the (N=XXX) in the table header. All decimal points should line up. If the minimum and maximum are output on one line as Minimum, Maximum then the comma should line up with the decimal point.
- If the original data has N decimal places, then the summary statistics should have the following decimal places:

Minimum and maximum: N Mean, median and CV%: N + 1

SD: N + 2



### Frequencies and percentages (n and %):

 Percent values should be reported inside parentheses, with one space between the count and the left parenthesis of the percentage. Parentheses should be justified to accept a maximum of 100.0 as a value and padded with blank space if the percent is less than 100.0. An example is given below: 77 (100.0%)

50 ( 64.9%)

0 (0.0%)

Percentages will be reported to one decimal place, except percents <100.0% but >99.9% will be presented as '>99.9%' (e.g., 99.99% is presented as >99.9%); and percents < 0.1% will be presented as '<0.1%' (e.g., 0.08% is presented as <0.1%). Rounding will be applied after the <0.1% and >99.9% rule. Eg ( <0.1%)</li>

(6.8%)

(>99.9%)

Percentages may be reported to 0 decimal places as appropriate (for example, where the denominator is relatively small).

• Where counts are zero, percentages of 0.0% should appear in the output.

### Confidence Intervals:

- As a rule confidence intervals are output to one place more than the raw data, and standard deviations and standard errors to two places more than the raw data
- Confidence intervals should be justified so that parentheses displayed on consecutive lines of a table "line up".
- Boundary values of confidence intervals should be separated by a comma.
- Boundary values should be padded as necessary to accept negative values and to allow alignment of the decimal place.
- An example is given below:

(-0.12, -0.10)

(9.54, 12.91)

### P-values:

• P-values should be reported to three decimal places, except values <1.000 but >0.999 will be presented as '>0.999' (e.g., 0.9998 is presented as >0.999); and values <0.001 will be presented as '<0.001' (e.g., 0.0009 is presented as <0.001). Rounding will be applied after the <0.001 and >0.999 rule

#### Ratios

• Ratios should be reported to one more decimal place than the original data.

### Spacing:

• There must be a minimum of 1 blank space between columns (preferably 2)



#### **Denominators:**

- If a different count other than the population count is used for a denominator (within the table) to calculate percentages, there should be a row in the table that identifies that number "n".
- Alternatively, a footnote should be included in each table with percentages to indicate the denominator for percentages.

#### Missing values

- A "0" should be used to indicate a zero frequency.
- A blank will be used to indicate missing data in an end-of-text table or subject listing.

#### FIGURE OUTPUT CONVENTIONS

- Figures should be provided in RTF files using the SAS Output Delivery System (ODS), as Computer Graphics Metafile (CGM) formatted graphical output generated by SAS.
- The CGM file itself should contain the title or footer.
- The image should be clear and of high quality when viewed in the Word document, and when printed.
- In general, boxes around the figures should be used.

#### **FOOTNOTE INFORMATION**

Footers should be defined as follows:

- A continuous line of underscores ('\_') will follow the body of the table or listing prior to any footnotes at the bottom of the page
- Table footnotes should be defined using compute statements in the proc report, and should appear directly after the body of the table
- The program path and name and version number (if applicable) should appear as footnote 1 at the bottom of the page
- The date/time stamp should appear as footnote 2 at the bottom of the page
- Footnotes should be left-aligned.
- Footnotes should be in sentence case.
- Only "typewriter" symbols are permitted eg "\*", "\$", "#", "@", "&" and "+".
- The choice of footnote symbols should be consistent. E.g. if you have the footnote "# indicates last observation carried forward" for one table, the same symbol and footnote should indicate LOCF for all tables.
- If text wraps across more than one line (for a note), the first letter for all lines of text after the first one will be indented to align beneath the first letter of the text in the first line.
- The page identification in the format Page X of Y (where Y is the total number of pages for the output) should appear in the first footnote, right aligned

Ordering of footnotes should be as follows:

1.) Source data listing reference, if necessary



- 2.) Abbreviations and definitions
- 3.) Formulae
- 4.) P-value significance footnote
- 5.) Symbols
- 6.) Specific notes
- Common notes from table to table should appear in the same order.
- The symbols should appear in the same order as what they are defined in the table or listing, from left to right.

#### PROGRAMMING INSTRUCTIONS

Programming instructions must appear in blue font at the end of each table or listing shell. Programming instructions, where necessary, should follow the table or listing shells in blue font, beginning with the words "Programming Note" followed by a colon. These include notes on the output, reminders of how to handle missing values, repeat shells for similar tables etc.

**Dates & Times** 

Depending on data available, dates and times will take the form yyyy-mm-ddThh:mm:ss.

**Presentation of Treatment Groups** 

For outputs, treatment groups will be represented as follows and in that order:

| Treatment<br>Group | For Tables and Graphs | For Listings |
|--------------------------|-----------------------|-----------------------|
| Placebo | Placebo | Placebo |
| Bempedoic Acid<br>180 mg | Bempedoic Acid 180 mg | Bempedoic Acid 180 mg |
| Not Randomized | Not Randomized | Not Randomized |

Presentation of Visits

For outputs, visits will be represented as follows and in that order:

| Long Name (default) | Short Name |
|---------------------|------------|
| Week -5 (Visit S1) | W-5 (VS1) |
| Week -4 (Visit S2) | W-4 (VS2) |
| Week -1 (Visit S3) | W-2 (VS3) |




| Long Name (default) | Short Name |
|---------------------|------------|
| Week 0 (Visit T1) | W0 (VT1) |
| Week 4 (Visit T2) | W4 (VT2) |
| Week 8 (Visit T3) | W8 (VT3) |
| Week 12 (Visit T4) | W12 (VT4) |
| Week 24 (Visit T5) | W24 (VT5) |

#### Listings

All listings will be ordered by the following (unless otherwise indicated in the template):

- randomized treatment
- center-subject ID,
- date (where applicable),
- For listings where non-randomized subjects are included, these will appear in a category after the randomized treatment groups labeled 'Not Randomized'.




# **APPENDIX 2. PARTIAL DATE CONVENTIONS**

Imputed dates will NOT be presented in the listings.

Algorithm for Treatment Emergence of Adverse Events:

| START DATE | ACTION |
|---|---|
| Known and | If AEPRIOR=Y then not TEAE |
| AESTART=study med | If AEPRIOR=N then TEAE |
| start date | |
| Known and AESTART>or | If start date < study med start date, then not TEAE |
| < study med start date | If start date > study med start date and <=study med |
| | end date + 30 , then TEAE |
| Partial | If AEPRIOR=Y then not TEAE |
| | Otherwise, |
| | If Impute 1 <sup>st</sup> of month if date is missing; impute 1 <sup>st</sup> of |
| | Jan if both date and month are missing. |
| | If resulting imputed start date is prior to study med |
| | start date, set as study med start date. If imputed |
| | start date is <= study med end date + 30 days, then |
| | TEAE; otherwise NOT TEAE |
| Missing | If AEPRIOR=Y then not TEAE |
| | Otherwise, |
| | Assumed TEAE |

Algorithm for Prior / Concomitant Medications:

Please note that the study med start date is the double-blind med start date.

| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| Known | Known | If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post study |



| START<br>DATE | STOP<br>DATE | ACTION |
|---|---|---|
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |
| | Missing | If stop date is missing could never be assumed a prior medication If start date <= end of treatment, assign as concomitant If start date > end of treatment, assign as post treatment |
| Partial | Known | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |
| | Partial | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown) and impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date and start date <= end of treatment, assign as concomitant If stop date >= study med start date and start date > end of treatment, assign as post treatment |
| | Missing | Impute start date as earliest possible date (i.e. first day of month if day unknown or 1st January if day and month are unknown), then: If stop date is missing could never be assumed a prior medication If start date <= end of treatment, assign as concomitant If start date > end of treatment, assign as post treatment |
| Missing | Known | If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'post treatment' |
| | Partial | Impute stop date as latest possible date (i.e. last day of month if day unknown or 31st December if day and month are unknown), then: If stop date < study med start date, assign as prior If stop date >= study med start date, assign as concomitant Cannot be assigned as 'post treatment' |



ESPERION THERAPEUTICS, INC. STATISTICAL ANALYSIS PLAN: PROTOCOL 1002-046 

| START<br>DATE | STOP<br>DATE | ACTION |
|---------------|--------------|-----------------------|
| | Missing | Assign as concomitant |




# APPENDIX 3. LIST OF DMC TABLES, LISTINGS AND FIGURES

# **TABLES**

| 14.1.1.1 | Patient Disposition – All Patients |
|---|---|
| 14.1.2.1a | Demographic and Other Baseline Characteristics – Full Analysis Set |
| 14.1.3.1 | Medical/Surgical History – Full Analysis Set |
| 14.1.3.3 | Targeted Cardiovascular History/Risk Factors – Full Analysis Set |
| 14.1.5.1 | Study Drug Compliance – Safety Analysis Set |
| 14.3.1.1 | Overview of Treatment-Emergent Adverse Events – Safety Analysis Set |
| 14.3.1.2 | Treatment-Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.3 | Serious Treatment-Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.4 | Related Treatment-Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.5 | Related Serious Treatment-Emergent Adverse Events by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.6 | Treatment-Emergent Adverse Events That Led to Discontinuation of Study Drug by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.8 | Treatment-Emergent AESIs by Maximum Severity, System Organ Class and Preferred Term – Safety Analysis Set |
| 14.3.1.15 | Investigator-reported Major Cardiac Events (MACE) by Event Type – Safety Analysis Set |
| 14.3.1.16 | Adjudicated Major Cardiac Events (MACE) by Event Type – Safety Analysis Set |
| 14.3.2.8 | Laboratory Parameters of Interest: Observed and Change from Baseline – Safety Analysis Set |
| 14.3.2.9 | Laboratory Parameters of Interest: Laboratory Abnormalities – Safety Analysis Set |




**QUINTILES** 

14.3.2.10 Quantitative Clinical Laboratory Evaluations: Lipids – Safety Analysis Set (note that this table is produced for DMC only)

## **FIGURES**

- 14.3.1 Boxplots of Hematology Parameters
- 14.3.2 Boxplots of Chemistry Parameters

The next 2 listings will created at the same time frame as DMC TLFs above. However, these 2 listings will be sent to Esperion Team only for monitoring thresholds for protocol deviations and for evaluable patients, but not sent to DMC members.

- Listing 16.2.3 Patient Inclusion per Analysis Population All Screened Patients
- Listing 16.2.4 Screen Failures All Screened Patients (note that this listing is produced for DMC only)




## **APPENDIX 4.** DETAILS OF MULTIPLE IMPUTATION METHOD

Missing Week 12 values will be imputed based on baseline values. The following table details the possible cohorts and which cohorts will be used for imputation. Missing Week 24 values will be imputed in the same way.

| | | | On | |
|---|---|---|---|---|
| | | Week 12 | Treatment | |
| | Treatment | Value | at Week 12 | Imputation Cohort(s) |
| | | | | Cohort 5: |
| | | | | Placebo patients with non-missing |
| 1 | Placebo | Missing | Yes | Week 12 |
| | | | | Cohorts 6 and 8 |
| 2 | BA | Missing | Yes | BA patients with non-missing Week 12 |
| | | | | Cohort 5: |
| | | | | Placebo patients with non-missing |
| 3 | placebo | Missing | No | Week 12 |
| | | | | Cohorts 5 and 7 |
| | | | | Placebo patients with non-missing Week 12 and not on |
| 4 | BA | Missing | No | treatment |
| 5 | placebo | Non-missing | Yes | |
| | D.4 | 3.7 | 3.7 | |
| 6 | BA | Non-missing | Yes | |
| 7 | placebo | Non-missing | No | |
| | piacebo | Non-missing | 100 | |
| 8 | BA | Non-missing | No | |

#### Imputation code for Cohorts 1-3.

proc mi; where cohort in(1,2,3,5,6,8); class trt01pn strata; monotone regression; var trt01pn strata base aval; run;

## Imputation code for Cohort 4.

proc mi; where cohort in(4,5,7); class strata; monotone regression; var base strata aval; run;



Two hundred imputed datasets will be created, with results from the analysis of each imputed dataset (ANCOVA) combined using Rubin's method.

## **APPENDIX 5. LIST OF ADVERSE EVENTS OF SPECIAL INTEREST**

| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|---|---|
| Creatine kinase elevations | Blood creatine phosphokinase abnormal |
| Creatine kinase elevations | Blood creatine phosphokinase increased |
| | Blood creatine phosphokinase MM |
| Creatine kinase elevations | abnormal |
| | Blood creatine phosphokinase MM |
| Creatine kinase elevations | increased |
| New onset or worsening diabetes mellitus | Blood glucose abnormal |
| New onset or worsening diabetes mellitus | Blood glucose increased |
| New onset or worsening diabetes mellitus | Diabetes mellitus |
| New onset or worsening diabetes mellitus | Diabetes mellitus inadequate control |
| New onset or worsening diabetes mellitus | Diabetic ketoacidosis |
| New onset or worsening diabetes mellitus | Glucose tolerance impaired |
| New onset or worsening diabetes mellitus | Glucose urine present |
| New onset or worsening diabetes mellitus | Glycosuria |
| New onset or worsening diabetes mellitus | Glycosylated haemoglobin increased |
| New onset or worsening diabetes mellitus | Hyperglycaemia |
| New onset or worsening diabetes mellitus | Impaired fasting glucose |
| New onset or worsening diabetes mellitus | Ketoacidosis |
| New onset or worsening diabetes mellitus | Ketosuria |
| New onset or worsening diabetes mellitus | Ketosis |
| New onset or worsening diabetes mellitus | Type 2 diabetes mellitus |
| New onset or worsening diabetes mellitus | Urine ketone body present |
| Hepatic disorders | Alanine aminotransferase abnormal |
| Hepatic disorders | Alanine aminotransferase increased |
| Hepatic disorders | Aspartate aminotransferase abnormal |
| Hepatic disorders | Aspartate aminotransferase abnormal |
| Hepatic disorders | Blood bilirubin abnormal |
| Hepatic disorders | Blood bilirubin increased |
| Hepatic disorders | Hepatic enzyme abnormal |
| Hepatic disorders | Hepatic enzyme increased |



| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|-------------------------------------|-----------------------------------|
| Hepatic disorders | Hypertransaminaseaemia |
| Hepatic disorders | Liver function test abnormal |
| Hepatic disorders | Liver function test increased |
| Hepatic disorders | Transaminases abnormal |
| Hepatic disorders | Transaminases increased |
| Hypoglycemia | Blood glucose abnormal |
| Hypoglycemia | Blood glucose decreased |
| Hypoglycemia | Hypoglycaemia |
| Hypoglycemia | Hypoglycaemic coma |
| Hypoglycemia | Hypoglycaemic encephalopathy |
| Hypoglycemia | Hypoglycaemic seizure |
| Hypoglycemia | Shock hypoglycaemic |
| Metabolic acidosis | Metabolic acidosis |
| Muscular disorders | Muscular weakness |
| Muscular disorders | Muscle necrosis |
| Muscular disorders | Muscle spasms |
| Muscular disorders | Myalgia |
| Muscular disorders | Myoglobin blood increased |
| Muscular disorders | Myoglobin blood present |
| Muscular disorders | Myoglobin urine present |
| Muscular disorders | Myoglobinaemia |
| Muscular disorders | Myoglininuria |
| Muscular disorders | Myopathy |
| Muscular disorders | Myopathy toxic |
| Muscular disorders | Necrotizing myositis |
| Muscular disorders | Pain in extremity |
| Muscular disorders | Rhabdomyolysis |
| Neurocognitive/Neurologic disorders | Amnesia |
| Neurocognitive/Neurologic disorders | Cognitive disorder |
| Neurocognitive/Neurologic disorders | Confusional state |
| Neurocognitive/Neurologic disorders | Disorientation |
| Neurocognitive/Neurologic disorders | Memory impairment |
| Neurocognitive/Neurologic disorders | Mental status changes |
| Renal disorders | Acute kidney injury |
| Renal disorders | Acute prerenal failure |
| Renal disorders | Blood creatinine abnormal |




| Adverse Event Terms per Protocol | Associated MedDRA Preferred Terms |
|---|---|
| Renal disorders | Blood creatinine increased |
| Renal disorders | Blood urea abnormal |
| Renal disorders | Blood urea increased |
| Renal disorders | Blood urea nitrogen/Creatinine ratio increased |
| Renal disorders | Creatinine renal clearance abnormal |
| Renal disorders | Creatinine renal clearance decreased |
| Renal disorders | Glomerular filtration rate abnormal |
| Renal disorders | Glomerular filtration rate decreased |
| Renal disorders | Gout |
| Renal disorders | Oliguria |
| Renal disorders | Prerenal failure |
| Renal disorders | Renal failure |
| Renal disorders | Renal function test abnormal |
| Renal disorders | Renal impairment |

## Addendum to Statistical Analysis Plan

Title: A RANDOMIZED, DOUBLE-BLIND, PARALLEL GROUP,

MULTICENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF BEMPEDOIC ACID (ETC-1002) 180 MG COMPARED TO PLACEBO ADDED TO BACKGROUND LIPID-MODIFYING THERAPY IN PATIENTS WITH ELEVATED LDL-

C WHO ARE STATIN INTOLERANT

**Protocol:** ETC-1002-046

Clinical Phase: 3

**Product:** ETC-1002 **Date:** Dec 18, 2018

Confidential Page 1 of 2


# Addendum to the Statistical Analysis Plan for Study 1002-046

## **Post-hoc Analyses**

Esperion completed the planned analysis as described in Study 1002-046 SAP for all data collected in the study.

After unblinding, some issues of clinical interest were identified. To address these issues, post-hoc analyses were performed to summarize the following: statin related adverse events prior to study entry, patients experiencing repeated and confirmed abnormal liver function tests after randomization, and percent change from baseline in LDL-C over time by background lipid modifying therapy (LMT). Finally, a sensitivity analysis was performed for the primary endpoint with Site 1020 excluded, since this was closed prematurely based on administrative and site accessibility issues.

The listing of tables for the post-hoc analyses is provided in the table below.

## Listing of new Tables for Study 1002-046.

| Table 17.1.1.1 | Statin Related Adverse Effect/ Full Analysis Set |
|---|---|
| Table 17.2.1.1 | Primary Efficacy Post-hoc Analysis: Percent Change from Baseline in Low Density Lipoprotein Cholesterol (LDL-C)/ |
| | Excluding Site 1021/ |
| | Full Analysis Set |
| Table 17.3.1.1 | Primary Efficacy Post-hoc Analysis: Percent Change from Baseline in Low Density Lipoprotein Cholesterol (LDL-C)/ |
| | By Background Lipid Modifying Therapy Lipid Modifying Treatment Subgroup/ |
| | Observed Data/ |
| | Full Analysis Set |
| Table 17.4.1.1 | Primary Efficacy Post-hoc Analysis: Percent Change from Baseline in Low Density Lipoprotein Cholesterol (LDL-C)/ |
| | By Background Lipid Modifying Therapy Lipid Modifying Treatment Subgroup/ |
| | On-Treatment Analysis/ |
| | Full Analysis Set |
| Table 17.5.1.1 | Post-Randomization Abnormal Liver Function Summary/ |
| | Safety Analysis Set |

Confidential Page 2 of 2